CLINICAL TRIAL: NCT03988712
Title: Establishing Absolute Iron Deficiency Anaemia Before Referring Patients to Colorectal Fast Track Clinics Can Help to Increase the Diagnostic Yield of the Bowel Cancer Screening Programme.
Brief Title: Measures to Increase the Effectiveness of Fast Track Colorectal Clinics for Iron Deficiency Anaemia.
Status: Completed | Type: Observational
Sponsor: Wirral University Teaching Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Mr Talal Majeed, Research Fellow, Wirral University Teaching Hospital NHS Trust
Other Study IDs: 161130
Record Dates: First submitted 2019-06-06; First posted 2019-06-17 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Cancer
Keywords: Anaemia; colorectal cancer; Iron deficiency anaemia
MeSH Terms: conditions — Colorectal Neoplasms; Anemia; Anemia, Iron-Deficiency | interventions — Colonoscopy; Gastroscopy; Colonography, Computed Tomographic; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Iron deficiency anaemia with bowel symptoms: Patients with IDA presenting with bowel symptoms like change in bowel habits, weight loss and abdominal mass other than rectal bleed
  Interventions: Diagnostic Test: Colonoscopy, gastroscopy, virtual colonoscopy, CT scan
- Iron deficiency anaemia with no bowel symptoms: Patients with IDA with no bowel symptoms
  Interventions: Diagnostic Test: Colonoscopy, gastroscopy, virtual colonoscopy, CT scan
- Iron deficiency anaemia with rectal bleeding: Patients with IDA and rectal bleeding
  Interventions: Diagnostic Test: Colonoscopy, gastroscopy, virtual colonoscopy, CT scan

INTERVENTIONS:
Diagnostic Test: Colonoscopy, gastroscopy, virtual colonoscopy, CT scan — Patients referred with a suspected bowel malignancy were subjected to top and bottom endoscopic examination or a cross sectional imaging like CT scan and MRI scan.

SUMMARY:
A retrospective cohort study was conducted from 2016-18 in a single busy district general hospital providing services to a population of 700,000 people.

In the study, patients with true IDA (low MCV and ferritin) were found to be more likely to have Colorectal cancer compared to any other type of anaemia which confirmed the latest guidelines for management of IDA. Compared to symptoms, only the presence of a mass on abdominal examination and rectal examination was found to be more likely associated with cancer.

DETAILED DESCRIPTION:
Although there are strict and specific guidelines for referring patients with iron deficiency anaemia (IDA) to fast track colorectal cancer (FT CRC) clinics for further assessment and investigation, patients with other types of anaemia are still referred by primary care physicians in the UK. Investigators aim was to find out whether this practice is correct, or if it is causing an overburden on colorectal clinics and endoscopy services. Investigators also want to find out whether true/absolute IDA has a higher predictive value for diagnosing colorectal cancer (CRC) compared to other types of anaemia and specific bowel symptoms.

Investigator's hypothesis was that patients with IDA are more likely to have CRC compared to patients with no anaemia or non-IDA anaemia. By confirming this hypothesis, Investigators can identify high risk patients from the population who can then be preferentially subjected to investigations mandated by guidelines. This strategy can help to increase the diagnostic yield of FT CRC clinics.

A retrospective cohort study was conducted from 2016-18 in a single busy district general hospital providing services to a population of 700,000 people.

In the study, patients with true IDA (low MCV and ferritin) were found to be more likely to have CRC compared to any other type of anaemia which confirmed the latest guidelines for management of IDA. Compared to symptoms, only the presence of a mass on abdominal examination and rectal examination was found to be more likely associated with cancer.

Physicians should be able to stratify patients based on blood indices when referring them to FT CRC clinics. Diagnostic yield of these clinics can be increased if clinicians strictly adhere to fast track guidelines and confirm true IDA before referring patients to clinic.

ELIGIBILITY:
Inclusion Criteria:

- Patients with age more than 18 years Presenting to fast track colorectal clinic

1. With bowel symptoms
2. Presenting with anaemia
3. Rectal bleeding

Exclusion Criteria:

* Any patient presenting through routine colorectal clinics

  1. With bowel symptoms
  2. Presenting with anaemia
  3. Rectal bleeding Aged less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective observational study from a busy district general hospital. A retrospective analysis of prospectively maintained data for FT CRC was performed. Data was selected from 2016-18. A cohort of 4177 patients presented to FT clinics. Among them 950 (22.74%) patients were referred with anaemia
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of colorectal cancer | 2 weeks
  diagnostic yield of colorectal cancer in patients presenting to fast track clinics with symptomatic ,asymptomatic anaemia, anaemia with normal blood indices, anaemia with Iron deficiency anaemia and certain bowel symptoms was measured. Patients were subjected to endoscopy for diagnosis. Diagnostic yield was expressed as diagnostic odds ratio and measured by statistical tools like Mantel Haenszel trend test and results are illustrated in the from of odds ratio. Crude odds ratio could not be used as association of binary outcome (colorectal caner or no cancer) with binary predictors in multiple case control groups was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: TALAL MAJEED, MRCS, Principal Investigator — Mr Talal Majeed
Locations (1):
- York Hospital, York, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
I have an excel sheet of the data and statistics done on the data which can be provided on request